CLINICAL TRIAL: NCT02471625
Title: Traumatic Brain Injury (TBI) Feasibility Study to Determine Possible Prognostic Indicators as Provided by the EPIC ClearView™
Brief Title: Traumatic Brain Injury Feasibility Study (EPIC-011)
Acronym: TBI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Epic Research & Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EPIC-011
Record Dates: First submitted 2015-06-04; First posted 2015-06-15 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Traumatic Brain Injury; Controls
Keywords: Controls
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Traumatic Brain Injury: Men and women ages 18-65 with suspected acute head trauma within 24-72hrs. of presentation, scoring a 3-15 on initial evaluation on GCS scale.
- Control: Men and women ages 18-65 with no history of head trauma and a score of 15 on the GCS scale.
  Interventions: Device: ClearView Scanning

INTERVENTIONS:
Device: ClearView Scanning
  Groups: Control

SUMMARY:
The purpose of this research study is to evaluate whether data made by the ClearView System can be used to detect whether someone has a traumatic brain injury and how severe the injury is.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a significant cause of death and disability in the U.S. The severity of a TBI may range from "mild" (i.e. a brief change in mental status or consciousness) to "severe" (i.e. an extended period of unconsciousness or memory loss after the injury). However, most TBI's that occur each year are mild and are commonly called concussions. Unfortunately, TBI terminology does not adequately describe the injury or impairment, its treatment, or the resulting outcomes. Due to the complexity of the human brain, each person's physiology can result in different patterns of impairment and secondary conditions, requiring different treatment or rehabilitation. The intent of EPIC ClearView™ TBI Feasibility (EPIC-011) is to collect data to further develop the ClearView™ Response Scale to measure electrophysiology associated with TBI

ELIGIBILITY:
Inclusion Criteria:

Suspected TBI population:

1. Acute head trauma within 24-72 hours of presentation
2. 18-65 age inclusive
3. GCS of 3-15 on initial evaluation in ED

Control population:

1. 18-65 age inclusive
2. GCS score of 15

Exclusion Criteria:

1. Current neurological disease
2. Current severe psychological disorder
3. History of substance or alcohol abuse
4. Under drug or alcohol influence, if so, must wait at least 24 hrs. prior to consent
5. Documented current diagnosis/treatment of cancer (including Sickle Cell Disease)
6. Current treatment to the head/brain (radiation, whole brain therapy, gamma knife)
7. Head injury in the last two years
8. Unwilling to sign informed consent
9. Pregnant or potentially pregnant
10. Pacemaker, automatic implanted cardiac defibrillator or other implanted electrical device
11. Connected to an electronic device that cannot be removed
12. Missing all or part of fingers or cuts/burns on pads of fingers
13. Long fingernails and unwilling to cut them and keep them cut for the duration of the study
14. Hand tremors or involuntary oscillations ("shaking") of the hands that prevents clear imaging

Additional exclusion criteria for control population:

Previous head trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women ages 18-65 who present to the ER with suspected head trauma and meet all inclusion and no exclusion criteria will be approached for consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Agreement of ClearView Scan versus Active Diagnosis | I day unless TBI population chooses to participate in one week follow up
  The EPIC ClearView software produces a Response Scale report that summaries the electrophysiological measurements associated with organ systems. The autonomic numbers indicate how the person's stress response is affecting different body systems and the physical numbers reflect physiological function. These measurements will then be compared to TBI diagnosis, based on one or two possible scans

SECONDARY OUTCOMES:
Comparison of TBI subjects to Controls | 1 day unless TBI population chooses to participate in one week follow up
  Will measure comparisons of data from one visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States